CLINICAL TRIAL: NCT02725736
Title: Tocolytic Therapy for Preterm Labor in Multiple Gestation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 755-15-TLV
Record Dates: First submitted 2016-03-22; First posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Labor Preterm Multiple
MeSH Terms: interventions — atosiban; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atosiban (Experimental): Women with twin pregnancy with preterm labor between 24 weeks 0 days and 32 weeks 6 days of gestation will be included and randomly assigned to the Atosiban group.
  Interventions: Drug: Atosiban
- Nifedipine (Experimental): Women with twin pregnancy with preterm labor between 24 weeks 0 days and 32 weeks 6 days of gestation will be included and randomly assigned to the Nifedipine group.
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Atosiban — After random allocation to a treatment group, women will receive Atosiban as follows:
  Atosiban was given as a single loading intravenous dose, 6.75 mg in 0.9% sodium chloride solution, followed by an intravenous infusion of 300 micrograms/min in 0.9% sodium chloride solution for the first 3 hours and then 100 micrograms/min for another 45 hours. The choice of the dose regimen for Atosiban was consistent with the recommendations of the product labeling.
  Arms: Atosiban
Drug: Nifedipine — After random allocation to a treatment group, women will receive Nifedipine as follows:
  Nifedipine was given as a loading dose of 20 mg orally followed by another two doses of 20 mg, 20-30 minutes apart as needed. Maintenance was started after 6 hours with 20-40 mg four times a day for a total of 48 hours.
  Arms: Nifedipine

SUMMARY:
To compare the tocolytic efficacy oxytocin receptor antagonist (Atosiban) with that of calcium channel blockers (Nifedipine) among women with multiple gestation who present with threatened preterm labor.

DETAILED DESCRIPTION:
Preterm birth remains the principal cause of early neonatal death. Infants born preterm (before 37 weeks' gestation) often suffer significant immediate morbidity and need lengthy stays in neonatal intensive care units. Moreover, there is a significant risk of long-term neurological morbidity in a proportion of the survivors. Patients with a multiple gestation are at significant risk for preterm labor and delivery as approximately 60% of all those pregnancies will be delivered preterm.

A number of oxytocin receptor antagonists have been developed, and of these, three, atosiban, barusiban and retosiban have been investigated in humans as tocolytic agents. To date, only atosiban is in use outside of clinical trials. Atosiban is an oxytocin receptor antagonist which was specifically developed for the treatment of preterm labor. Early reports of the use of Atosiban for tocolysis showed promise both in vitro and in animal studies, and preliminary studies in pregnant and non-pregnant humans suggested a very low incidence of maternal side effects .

ELIGIBILITY:
Inclusion Criteria:

1. Twin pregnancy
2. Gestational age between 24+0 and 32+6 weeks
3. Intact amniotic membranes
4. Threatened preterm labor
5. Age 18-50.

Exclusion Criteria:

1. Rupture of membranes
2. Vaginal bleeding resulting from placenta previa or placental abruption
3. Fever above 38°C
4. Severe preeclampsia
5. Maternal cardiovascular or liver diseases
6. Systolic blood pressure less than 90 mm Hg
7. Known uterine malformation
8. Intrauterine growth restriction below the fifth percentile
9. Non-reassuring fetal status
10. Antepartum diagnosis of major fetal malformations
11. Fetal death
12. Previous tocolytic therapy or Betamethasone treatment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Duration of labor | 48 hours

SECONDARY OUTCOMES:
Infant morbidity | 28 days
  Defined as the number of infant morbidity up to 28 days from birth.
Chronic lung disease | 28 days
  Defined as the number of participants with need for supplemental oxygen at 28 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Yariv Yogev, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046